CLINICAL TRIAL: NCT01503008
Title: Proteus Sustained Behavior Change Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Proteus Digital Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB-SBCT2DM
Record Dates: First submitted 2011-12-28; First posted 2012-01-02 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Sulfonylurea Compounds; Thiazolidinediones; Dipeptidyl-Peptidase IV Inhibitors; Glycoside Hydrolase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sustained Behavior Change system support (Experimental)
  Interventions: Device: Proteus Sustained Behavior Change system
- Control (Active Comparator)
  Interventions: Drug: Regularly prescribed diabetes medicines (metformin, sulfonylureas, thiazolidinediones, DPP-IV inhibitors, alpha-glucosidase inhibitors)

INTERVENTIONS:
Device: Proteus Sustained Behavior Change system — The SBC system uses ingestible and wearable sensing devices and mobile phones to reinforce positive behaviors around medication usage, exercise and rest. Subjects will be taking their regularly prescribed oral hypoglycemics (metformin, sulfonylureas, thiazolidinediones, DPP-IV inhibitors, alpha-glucosidase inhibitors); glucometer
  Arms: Sustained Behavior Change system support
Drug: Regularly prescribed diabetes medicines (metformin, sulfonylureas, thiazolidinediones, DPP-IV inhibitors, alpha-glucosidase inhibitors) — Oral hypoglycemics (metformin, sulfonylureas, thiazolidinediones, DPP-IV inhibitors, alpha-glucosidase inhibitors) at subjects' regularly prescribed doses; glucometer
  Arms: Control

SUMMARY:
The study will test whether the Proteus Sustained Behavior Change (SBC) System will help Type 2 diabetics feel more able to perform self-care activities, feel less distressed about diabetes, and reduce mean fasting blood glucose levels. The SBC system uses ingestible and wearable sensing devices and mobile phones to reinforce positive behaviors around medication usage, exercise and rest.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported diagnosis of Type 2 Diabetes Mellitus within the past 2-12 months
* Hemoglobin A1c ≥7.5 and ≤11, obtained with the point-of-care HbA1c diagnostic device during the enrollment visit
* Self-reported current use of metformin for Type 2 diabetes
* Male or female ≥ 18
* Outpatient
* Self-reported capacity to perform "moderate" exercise, as specified by in the 2010 joint American College of Sports Medicine/American Diabetes Association guidelines
* Designation of one caregiver to be involved in the study for its entire duration. A caregiver can be a relative, friend, or trained or untrained hired individual.
* Self-reported mobile phone reception at home and/or at work
* Willingness to adhere to study procedures, including troubleshooting of the Raisin System by a third-party if needed. The third party will be blinded to any personal subject identifiers.
* Capacity to read and speak English proficiently, as judged by the investigator during the screening interview
* Capacity to understand the instructions for the study, as judged by the investigator during the screening interview

Exclusion Criteria:

* Self-reported treatment with metformin for less than 2 months at the time of screening
* Self-reported adverse reaction to metformin (e.g., ongoing nausea, vomiting, bloating, diarrhea) or to other concomitant medications being administered at the time of screening
* Self-reported use of injectable hypoglycemic agents, such as insulin, exenatide, liraglutide or pramlintide
* Physical or medical condition that could prevent safe participation in moderate levels of physical activity, as surveyed by the Physical Activity Readiness Questionnaire (PAR-Q) and interpreted by the investigator
* Inability to use a mobile phone (e.g., to find icons or to open and to read a SMS), or inability to operate the approved glucometer that will be provided for use in the study
* Self-reported current (i.e., in the last 12 months) alcohol or drug abuse (including, but not limited, to use of marijuana)
* Positive urine pregnancy test for women
* Women of child bearing potential who are not using a medically accepted means of contraception. Accepted means of contraception include oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or partner with vasectomy
* Self-reported history of myocardial infarction within past 60 days
* Self-reported history of cerebral vascular accident within past 60 days
* Self-reported history of skin sensitivity to adhesive medical tape or metals
* Self-reported history of acute or chronic dermatitis, excluding atopic dermatitis
* Self-reported allergies that could preclude safe participation in the study
* Current participation in another clinical study, or participation in a clinical study in the past 30 days during which an investigational device or drug was used
* Any condition that, in the investigator's opinion, would preclude the subject's being able to meet all of the protocol requirements, or would compromise the subject's safety during participation in the study
* Presence of cognitive impairment, as judged by the investigator during the screening interview
* Inability to provide informed consent for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy | 3 months
  As measured by the 13-item self-efficacy expectancies and outcomes expectancies sub-scale of the Multidimensional Diabetes Questionnaire

SECONDARY OUTCOMES:
Perceived effectiveness of caregiver support | 3 months
  As measured by the 12-item positive reinforcing behaviors and misguided support sub-scale of the Multidimensional Diabetes Questionnaire
Diabetes-related distress | 3 months
  As measured by the 20-item Problem Areas In Diabetes scale
At-home measurements of fasting glucose | 1, 6, 12 weeks
  Weekly average for each time point
In-clinic measurements of fasting glucose | 0, 6, 12 weeks
  Discrete lab measurement
Usability | 3 months
Device-related and -unrelated adverse events | Up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Jethwani, MD, Principal Investigator — Center for Connected Health, Partners Healthcare; Michael J Coons, PhD, Principal Investigator — Northwestern University; Bonnie Spring, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Center for Connected Health, Partners Healthcare, Boston, Massachusetts